CLINICAL TRIAL: NCT03201614
Title: Comparative Evaluation of the Performance and Safety of A-CP HA Kit, for the Preparation of a Combination of Platelet Rich Plasma and Hyaluronic Acid, Versus Hyaluronic Acid Alone and Placebo in Patients With Knee Osteoarthritis
Brief Title: Comparative Evaluation of A-CP HA Kit, Hyaluronic Acid and Placebo for the Treatment of Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regen Lab SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RL 04
Record Dates: First submitted 2017-06-26; First posted 2017-06-28 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Knee Osteoarthritis
Keywords: platelet-rich plasma, hyaluronic acid, knee osteroarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- A-CP HA (Experimental): Patients randomized in this group will be treated with a combination of platelet-rich plasma plus hyaluronic acid prepared with A-CP HA Kit.
  Interventions: Device: A-CP HA Kit
- ArthroVisc 40 (Active Comparator): Patients randomized in this group will be treated with hyaluronic acid only (ArthroVisc 40); hyaluronic acid is the same as the one contained in the A-CP HA Kit.
  Interventions: Device: ArthroVisc 40
- Placebo (Placebo Comparator): Patients randomized in this group will be treated with a saline solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Device: A-CP HA Kit — Patients randomized in this group will receive two injections of platelet-rich plasma/hyaluronic acid prepared with the A-CP HA Kit at Day 0 and Month 2
  Arms: A-CP HA
Device: ArthroVisc 40 — Patients randomized in this group will receive two injections of hyaluronic acid only (ArthroVisc 40) at Day 0 and Month 2
  Arms: ArthroVisc 40
Drug: Placebo — Patients randomized in this group will receive two injections of a saline placebo at Day 0 and Month 2
  Arms: Placebo

SUMMARY:
Hyaluronic acid (HA) is a major component of synovial fluid, to which it confers viscosity and elasticity. It has been shown that the rheological properties of the synovial fluid decrease in patients with osteoarthritis. Intra-articular injections of hyaluronic acid represents a commonly used therapeutic option to relieve osteoarthritic symptoms, by exerting a mechanical action on cartilaginous structures of the joints, thus leading to reduced pain and improved joint function.

Platelet-rich Plasma is an autologous product prepared from the patient's own blood. Potential benefits of platelet-rich plasma for the treatment of cartilage defects have been suggested by many in vitro and animal studies. There are an increasing number of clinical studies assessing the benefits of platelet rich plasma in the treatment of osteoarthritis, showing that platelet rich plasma improves symptoms with no serious adverse events reported.

On the basis of the above, HA and platelet-rich plasma have the potential to provide added benefits in osteoarthritis symptoms when combined, in particular in patients who have had previous intra-articular HA treatment but who are still experiencing pain. Preliminary evidence to this effect was presented at the 2014 Annual Congress of the French Rheumatology Society by a group of French investigators. Renevier and Marc enrolled patients who had not experienced adequate symptom relief from previous intra-articular HA treatment and treated them with HA plus platelet-rich plasma prepared using A-CP HA Kit. Of the 71 patients treated, approximately 90% were classified as responders based on the OMERACT-OARSI criteria.

The A-CP HA Kit allows for the preparation of a homogenous solution of platelet-rich plasma and HA, intended to be injected intra-articularly for the treatment of pain in osteoarthritis. In patients who had previous intra-articular HA treatment but who are still experiencing pain, treatment with HA plus platelet rich plasma could provide a safe and reproducible option before surgery.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a degenerative disease of the joint cartilage. The evolution of this condition is characterized by the following symptoms: pain, joint cracking/popping, stiffness, deformity, loss of mobility and especially in the case of knee osteoarthritis, swelling (synovial effusion).

Osteoarthritis can lead to functional impairment and deformities thereby causing degradation of quality of life and may result in disabilities. Due to the fact that the knees and hips are weight bearing, osteoarthritis of these joints is often more disabling for persons who are affected by this condition.

Osteoarthritis is the most common joint disorder in the United States. Among adults 60 years of age or older, the prevalence of symptomatic knee osteoarthritis is approximately 10% in men and 13% in women. The number of people affected with symptomatic OA is likely to increase due to the aging of the population and the obesity epidemic.

A healthy joint is composed of two bone ends covered by cartilage (hyaline cartilage). This allows for shock absorption and for the bones to slide over one another with ease, thus ensuring the joint mobility. Synovial fluid (synovium) that surrounds the cartilage acts as lubrication and nutrition for the articular cartilage. It is mainly composed of hyaluronic acid, a glycosaminoglycan which binds to water molecules which in turn will result in a very viscous solution thereby giving the synovial fluid its shock absorbing properties. It has been shown that the rheological properties of synovial fluid decrease with age and in patients suffering from osteoarthritis, which may cause symptoms of pain and physical loss of function as seen in gonarthrosis, for example.

Osteoarthritis has multiple causative agents, many of which are not yet fully understood. However, a number of risk factors including age, gender, genetics, obesity, joint trauma, certain sports or professional activities are currently known. Conventionally, there is a distinction between so-called primary osteoarthritis, for which there is no obvious predisposition (of unknown origin) and secondary osteoarthritis, related to previous trauma or joint diseases. The secondary type represents the most common form of osteoarthritis.

There are many and varied possibilities for treating gonarthrosis which include both medicated and non-medicated routes. Among these, physical therapy and an improved life style (weight loss, use of suitable shoe inserts, regular physical activity etc.) are an essential component in the management of knee osteoarthritis.

In terms of medication, the administration of analgesics and non-steroidal anti-inflammatory drugs (NSAIDs) is the standard treatment. However, although they promptly act against pain and inflammation, they only have a limited effect over time in treating the symptoms without acting upon the cause.

Slow acting anti-rheumatic drugs, including glucosamine, chondroitin sulphate, diacerhein, soybean and avocado unsaponifiables on the contrary have a delayed action on the pain and joint function. Although still widely used in clinical practice for their chondroprotective effect, they have moderate efficacy and primarily allow for the reduction of analgesic and anti-inflammatory drug doses.

Corticoid infiltrations occupy an important place in the therapeutic range of osteoarthritis, especially when analgesics and anti-inflammatory drugs fail to relieve an inflammatory flare. The observed effect, however, has a limited effect over time.

Intra-articular injections of hyaluronic acid (viscosupplementation treatment) are currently the treatment of choice in gonarthrosis as they can relieve symptoms for several months at a time. These are designed to exert a mechanical action on cartilaginous structures of the joints, leading to a reduction in pain and improvement in the joint function. The effectiveness of hyaluronic acid is widely documented. Indeed, many clinical trials testing different hyaluronic acid preparations have been carried out in humans, some of which report results versus a saline placebo. Most of these studies conclude to the superiority of hyaluronic acid regardless of its molecular weight.

More recently, the injections of platelet rich plasma were found to be an attractive treatment option, due to the autologous nature of the product and its mechanism of action. Indeed, the action of platelet rich plasma is not based on sustainable viscoelasticity of the product, but on biological stimulation of mesenchymal stem cells (MSCs) and cartilaginous cells. Many in vitro studies have already demonstrated the effects of isolated growth factors on stimulation and chondrogenic differentiation of mesenchymal stem cells.

The clinical use of isolated growth factors is impossible today with regard to their mode of production and the potential risk to human health. The autologous platelet rich plasma is the simplest and safest solution to provide usable growth factors in a clinical setting. The interest and potential efficacy of platelet-rich plasma in the treatment of cartilage lesions have already been tested in vitro:

* Platelet-rich plasma increases the synthesis of proteoglycans and collagen in the extracellular matrix of cultured intervertebral disc cells
* Platelet-rich plasma stimulates the proliferation and biosynthesis of the matrix of articular chondrocytes in pigs
* Platelet-rich plasma increases the expression of the "cartilage oligomeric matrix protein" (COMP) Platelet-rich plasma was superior to a standard culture medium in the proliferation and differentiation of mesenchymal stem cells into chondrocytes At the clinical level, a number of studies showed improved symptoms with no serious adverse effects. When compared to hyaluronic acid injections, platelet-rich plasma treatment demonstrated superiority in terms of reduced pain, stiffness and function.

These results suggest that platelet-rich plasma, by its specific mechanism of action, is an effective and innovative tool in the therapeutic arsenal for the treatment of symptomatic gonarthrosis.

On the basis o the above, it is reasonable to assume that platelet-rich plasma and hyaluronic acid have the potential to provide added benefits in osteoarthritis when combined, in particular in patients who have had previous intra-articular HA treatment but who are still experiencing pain. Preliminary evidence to this effect was presented at the 2014 Annual Congress of the French Rheumatology Society by a group of French investigators. Renevier and Marc enrolled patients who had not experienced adequate symptom relief from previous intra-articular HA treatment and treated them with the combination of platelet rich plasma and HA prepared using A-CP HA Kit. Of the 71 patients treated approximately 90% were classified as responders based on the OMERACT-OARSI criteria.

The A-CP HA Kit, manufactured by Regen Lab SA, Le Mont-sur-Lausanne, VD, Switzerland, allows for the preparation of a homogenous solution of platelet-rich plasma and HA. The product is intended to be injected intra-articularly for the symptomatic treatment of pain. In patients who had previous intra-articular HA treatment but who are still experiencing pain, treatment with HA plus platelet-rich plasma could provide a safe and reproducible option before surgery.

The objective of this study is to investigate if a biological treatment based on a combination of platelet-rich plasma and hyaluronic acid obtained with A-CP HA Kit is statistically superior to HA alone, on one hand, and to a saline placebo, on the other hand, to reduce overall knee osteoarthritis symptoms, and particularly pain, and thus improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis grade 2-3 according to the Kellgren & Lawrence grading scale, as defined on knee radiographs (less than 3 months old: face view, schuss view, profile and patellar axial view at 30°)
* Knee Pain level of at least 3 on the 0-10-point WOMAC A subscale
* Bilateral osteoarthritis provided that the contralateral knee has a pain no more than 2 on the 0-10 point scale, and not requiring systemic analgesic treatment except paracetamol until the maximum dose of 4g per day

Exclusion Criteria:

* Grade <2 or >3 OA according to the Kellgren and Lawrence grading scale
* Bilateral osteoarthritis provided that the contralateral knee has a pain more than 2 on the 0-10 point scale and requiring systemic analgesic treatment or paracetamol more than 4g per day
* Viscosupplementation in the treatment site in the past 3 months
* Corticosteroid injection in the treatment site in the previous 3 months
* Systematic use of corticosteroid (except those that are inhaled) within 3 months
* History of allergy to hyaluronic acid
* Rheumatological disorders
* Clinical evidence of local inflammation such as redness or heat of the joint
* Current or medical history of autoimmune disease
* Surgery or arthroscopy surgery in the affected knee in the past 3 months
* Local infection in the affected knee
* Hematologic or clotting disorders (thrombocytopenia) or blood coagulation (deficit-blood dyscrasia)
* Anaemia (Haemoglobin < 10g/dl)
* Platelet count below 150/mmc
* Anticoagulant treatment
* Viral disease (hepatitis, herpes, varicella, zona, etc.)
* Renal failure or hemodialysis
* Acute infection
* Immunosuppressive states
* Malignant disease
* Recent fever (within previous 2 weeks) or serious disorders (liver disease, active gastroduodenal ulcer, digestive hemorrhage, etc.)
* Pregnancy or breastfeeding or planning pregnancy during the course of the study
* Immunosuppressants within the past 6 weeks or ongoing
* Uncontrolled diabetes
* Participation in another clinical study in the past 3 months
* Ongoing participation in another OA clinical study
* Fracture, skeletal dysplasia, congenital or acquired deformity that affects the knee
* Hemoglobin A1C > 8% within 8 weeks prior to the study treatment
* Have been given the diagnosis of fibromyalagia, neuropathic pain syndrome, or depression
* Refusal to sign or inability to give Informed Consent
* Inability to understand or comply with the requirements of the study
* Any other reason which may interfere with the proper conduct of the study, in the investigator's opinion

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Variation in overall OA-related symptoms | 6 Months
  It will be assessed by the mean difference in total WOMAC score on a 100-mm VAS between baseline and Month 6
Variation in pain at walking (WOMAC A1 score) | 6 Months
  II t will be assessed by the mean difference on a 100-mm VAS between baseline (D0) and Month 6

SECONDARY OUTCOMES:
Variation in overall OA-related symptoms, between baseline (D0) and Month 1 (D30), Month 2, Month 3, Month 4, and Month 12 | 12 Months
  It will be assessed by the mean difference in total WOMAC score on a 100-mm VAS between baseline (D0) and Month 1, Month 2, Month 3, Month 4, and month 12.
Variation in pain at walking (WOMAC A1 score), between baseline (D0) and Month 1 (Day 30), Month 2, Month 3, Month 4, and Month 12 | 12 Months
  It will be assessed by the mean difference in WOMAC A1 score on a 100-mm VAS between baseline (D0) and Month 1 (Day 30), Month 2, Month 3, Month 4, and Month 12
Variation of general pain, between baseline (D0) and Month 1 (Day 30), Month 2, Month 3, Month 4, Month 6 and Month 12 | 12 Months
  It will be assessed by the mean difference in total WOMAC A score on a 100-mm VAS between baseline (D0) and Month 1 (Day 30), Month 2, Month 3, Month 4, Month 6 and Month 12
Variation of joint stiffness, between baseline (D0) and Month 1 (Day 30), Month 2, Month 3, Month 4, Month 6 and Month 12 | 12 Months
  It will be assessed by the mean difference in total WOMAC B score on a 100-mm VAS between baseline (D0) and Month 1 (Day 30), Month 2, Month 3, Month 4, Month 6 and Month 12
Variation of joint function, between baseline (D0) and Month 1 (Day 30), Month 2, Month 3, Month 4, Month 6 and Month 12 | 12 Months
  It will be assessed by the mean difference in total WOMAC C score on a 100-mm VAS between baseline (D0) and Month 1 (Day 30), Month 2, Month 3, Month 4, Month 6 and Month 12
% of OMERACT-OARSI responders | 12 Months
  It will be assessed at Month 1, Month 2, Mont 3, Month 4, Month 6, and Month 12
Patient's global assessment on a 7-point scale | 12 Months
  It will be assessed at Month 1, Month 2, Mont 3, Month 4, Month 6, and Month 12
Patient's global assessment on a 7-point scale at Month 1 (D30), Month 2, Mont 3, Month 4, Month 6, and Month 12 Clinician's global assessment on a 7-point scale | 12 Months
  It will be assessed at Month 1, Month 2, Mont 3, Month 4, Month 6, and Month 12
Variation of the patient's quality of life | 12 months
  It will be assessed by the variation in the SF-36 questionnaire, between baseline (D0) and Month 1 (Day 30), Month 2, Month 3, Month 4, Month 6 and Month 12
Rescue medication | 12 Months
  Comparison of the use of rescue medication between the three groups of treatment at baseline, Month 1, Month 2, Month 3, Month 4, Month 6 and Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Bert Mandelbaum, MD, Principal Investigator — Santa Monica Orthopaedic & Sports Medicine Group; Nicholas Sgaglione, MD, Principal Investigator — Northwell Health
Locations (1):
- Bert Mandelbaum, MD, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided